CLINICAL TRIAL: NCT05966831
Title: A Randomized Effectiveness Trial of Metacognitive Self Control and Job Interview Training
Brief Title: Metacognitive Self Control and Job Interview Training
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not meet enrollment for analysis
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Matthew Smith, Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: HUM00234352
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Self-Control; Recidivism
Keywords: employment
MeSH Terms: conditions — Self-Control; Recidivism

STUDY DESIGN:
Intervention Model Description: Group 1 will receive two interventions: Metacognitive Self-Control Training plus Virtual Reality Job Interview Training.
  Group 2 will receive one intervention: Virtual Reality Job Interview Training
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metacognitive Self-Control Training (MCT) + Virtual Reality Job Interview Training (VR-JIT) (Experimental): This group will receive the MCT intervention plus the VR-JIT intervention. We are anticipating 6-8 weeks, with 1-3 sessions per week for each intervention.
  Interventions: Behavioral: Metacognitive Self-Control Training (MCT); Behavioral: Virtual Reality Job Interview Training (VR-JIT)
- Virtual Reality Job Interview Training (VR-JIT) (Experimental): This group will receive just the VR-JIT intervention. We are anticipating 6-8 weeks, with 1-3 sessions per week for this intervention.
  Interventions: Behavioral: Virtual Reality Job Interview Training (VR-JIT)

INTERVENTIONS:
Behavioral: Metacognitive Self-Control Training (MCT) — Metacognitive Self-Control Training (MCT) was originally developed by the Michigan Skills Project for students in middle/high school. The MCT training intervention has been updated to be suitable for adults. MCT is a lecture style intervention that encompasses 13 modules (over the course of 4 weeks) on improving self-control that is to be delivered in a community setting. Across the training, participants will learn new "tools" for improving self-control.
  Arms: Metacognitive Self-Control Training (MCT) + Virtual Reality Job Interview Training (VR-JIT)
Behavioral: Virtual Reality Job Interview Training (VR-JIT) — VR-JIT provides trainees with an opportunity to repeatedly practice interviewing for a job at fictional company 'Wondersmart'. Prior to interviewing, trainees review self-guided e-learning materials on how to find, prepare for, succeed in, and follow-up on job interviews that includes the review of 10 job interview skills. Trainees also complete an online job application for one of 14 jobs (e.g., cashier, clerical, customer service, food services, inventory, janitorial, web developer) that informs the virtual interview experience.

SUMMARY:
The study is a randomized controlled trial (RCT) that assesses the effectiveness of a metacognitive self-control training intervention (MCT) in conjunction with virtual-reality job interview training (VR-JIT) in a sample of formerly incarcerated individuals. The study also includes an implementation evaluation.

DETAILED DESCRIPTION:
The goal is to conduct a randomized controlled trial (RCT) that assesses the effectiveness of a metacognitive self-control training intervention (MCT) in conjunction with virtual-reality job interview training (VR-JIT) in a sample of formerly incarcerated individuals, as well as complete an implementation evaluation. Participants will be recruited who who: 1) have previously been incarcerated (e.g., jail, prison), 2) have reentered society, 3) 18 years of age or older, 4) currently are a part of the A Brighter Way program. A Brighter Way is a local re-entry program in Ypsilanti, Michigan (MI) that focuses on helping formerly incarcerated individuals (living in Washtenaw county) build stable and successful lives. Participants will be randomly assigned to conditions where they either receive both MCT and VR-JIT interventions, or where they receive an Active-Control Activity and VR-JIT intervention (with an allocation ratio of 1:1). To assess the effectiveness of MCT, researchers plan to compare behavioral and self-report measures of self-control pre and post interventions, as well as assess employment and recidivism outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Actively enrolled in A Brighter Way Program
* 3rd grade reading level or higher

Exclusion Criteria:

* Has uncorrected hearing or visual problem that prevents them from using the training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Self-Control Measured by Brief Self-Control Scale (BSCS) | Baseline and posttest (approximately 8 weeks after baseline)
  The measure is a Likert Scale style questionnaire. 13 items are scored from 1 (not at all) to 5 (Very much). The total score is calculated from adding all items together and higher scores indicate higher levels of self-control.
Change in Self-Control Measured by Barratt Impulsiveness Scale | Baseline and posttest (approximately 8 weeks after baseline)
  The measure is a Likert Scale style questionnaire. 30 items are scored from 1 (Rarely/Never) to 4 (Almost Always/Always). The total score is calculated from adding all items together and range from 30 to 120; higher scores indicate higher levels of impulsiveness.
Change in Self-Control Measured by Short Form Self-Regulation Questionnaire | Baseline and posttest (approximately 8 weeks after baseline)
  The measure is a Likert Scale style questionnaire. 31 items are scored from 1 (Strongly Disagree) to 5 (Strongly Agree). The total score is calculated from adding all items together. Higher scores indicate higher self-regulation capacity.
Change in Adult Attention Deficit/Hyperactivity Disorder (ADHD) Symptomology measured by ADHD Self-Report Scale (ASRS) | Baseline and posttest (approximately 8 weeks after baseline)
  The Adult ADHD Self-Report Scale (ASRS) is an instrument consisting of the eighteen Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision (DSM-IV TR) criteria. Six of the eighteen questions were found to be the most predictive of symptoms consistent with ADHD. These six questions are the basis for the ASRS v1.1 Screener and are also Part A of the Symptom Checklist. Part B of the Symptom Checklist contains the remaining twelve questions. All questions utilize a Likert scale from Never, Rarely, Sometimes, Often, to Very Often.
Change in Adult Attention Deficit/Hyperactivity Disorder (ADHD) Symptomology measured by the Structured Clinical Interview (SCID-RV) for The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) | Baseline and posttest (approximately 8 weeks after baseline)
  The Structured Clinical Interview (SCID-RV) for DSM-5 for Adult Attention-Deficit/Hyperactivity Disorder measures ADHD symptomology. The module is made up of 5 major criteria with items in each criteria using a 3 point Likert scale ranging from 1 "absent or False" to 3 "threshold or true". This module uses a dichotomous scoring method that indexes whether a symptom is present or not. Only responses of "threshold or true" are coded as symptom present, while responses of "subthreshold" or "absent or false" are coded as symptom absent, so each individual will have a score of symptom absent = 0, and symptom present = 1 for criteria A through E.
Change in Employment Outcome | Baseline and 9 Month Follow Up (9 Months after randomization)
  Employment survey indicating that participants are either employed (1) or unemployed (0).

SECONDARY OUTCOMES:
Change in Recidivism | Baseline and throughout 9 Month Follow Up (9 Months after randomization)
  Researchers will track if a participant becomes re-incarcerated throughout the entire study. This will be marked as Yes (1) or No (0) in our database tracking.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No